CLINICAL TRIAL: NCT04054570
Title: The Geneva Lake Study Update : An Overview of Home Non-Invasive Ventilation 15 Years Later
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Jean-Paul Janssens, Professor Jean-Paul Janssens, University Hospital, Geneva
Other Study IDs: n°PB_2016-00925/15-275
Record Dates: First submitted 2019-07-21; First posted 2019-08-13 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Home Non-Invasive Ventilation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adaptive servo-ventilation patients: All patients under adaptive servo-ventilation in the Geneva Lake area and details of the specifics indications, population treated and venitator settings
  Interventions: Other: No intervention
- Barometric and Volumetric patients: All patients under barometric and volumetric ventilation in the Geneva Lake area and details of the specifics indications, population treated and venitator settings
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No Intervention

SUMMARY:
A multicenter cross-sectional observational study was conducted in the counties of Geneva and Vaud (1'271'957 inhabitants in 2016 and 1'288'090 inhabitants in 2017 ) and included all subjects under home NIV followed by the two university hospitals of Geneva and Lausanne (HUG and CHUV), one private regional general hospital (La Tour Hospital), one pulmonary rehabilitation center (Rolle Hospital) and 38 pulmonologists in private practice (for a total of 43, 18 in Geneva and 20 in Vaud). In Switzerland home NIV can be prescribed, initiated and followed by a pulmonologist in private practice without referring to a hospital center. The coordinating institution for this project was the Geneva University Hospital (HUG).

The investigator's goals were to update the prevalence of home NIV, the description of the population involved, the devices used, their settings, compliance, and a large array of technical data to provide a complete photography of home NIV in an area with 30 years of experience in this field. We also aimed to collect data regarding pursuit or interruption of NIV and survival during observation period.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged over 18 years old undergoing long term home NIV for at least 3 months and living in the Cantons of Geneva or Vaud were eligible for the study.

Exclusion Criteria:

* The only exclusion criteria was invasive ventilation (tracheostomy).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all age undergoing long term home NIV for at least 3 months and living in the Cantons of Geneva or Vaud
Sampling Method: Non-Probability Sample
Enrollment: 947 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis | 01.06.2016-10.07.2018
  Diagnosis leading to NIV. 5 disease categories with identification of the percentage of patients with SRBD, COPD, Overlap syndrome, OHS, NMD, restrictive chest wall and lung disorders. All data were analyzed using descriptive statistics. Qualitative parameters were described as frequencies and percentages and quantitative parameters were described as mean and standard deviation (SD) or as median and interval interquartile (IQR). Comparisons between groups were performed using chi-square tests or Fisher exact tests for qualitative parameters and analysis of variance (one-way ANOVA) or Kruskal-Wallis tests for quantitative parameters, as appropriate.

SECONDARY OUTCOMES:
Baseline characteristics | 01.06.2016-10.07.2018
  Comorbidities, age, gender. All data were analyzed using descriptive statistics. Qualitative parameters were described as frequencies and percentages and quantitative parameters were described as mean and standard deviation (SD) or as median and interval interquartile (IQR). Comparisons between groups were performed using chi-square tests or Fisher exact tests for qualitative parameters and analysis of variance (one-way ANOVA) or Kruskal-Wallis tests for quantitative parameters, as appropriate.
Survival | 01.06.2016-01.05.2021
  Analyze short-term mortality rate and risk factors. All data were analyzed using descriptive statistics. Qualitative parameters were described as frequencies and percentages and quantitative parameters were described as mean and standard deviation (SD) or as median and interval interquartile (IQR). Comparisons between groups were performed using chi-square tests or Fisher exact tests for qualitative parameters and analysis of variance (one-way ANOVA) or Kruskal-Wallis tests for quantitative parameters, as appropriate.
Leaks | 01.06.2016-10.07.2018
  Investigate modifiable and non-modifiable risk factors asssociated with non intentional air leaks during home non invasive ventilation (NIV). Air leaks are identified by the built in software of the ventilator and clinicians download these data onto a computer. Leaks are expressed in ml or liters. All data were analyzed using descriptive statistics. Qualitative parameters were described as frequencies and percentages and quantitative parameters were described as mean and standard deviation (SD) or as median and interval interquartile (IQR). Comparisons between groups were performed using chi-square tests or Fisher exact tests for qualitative parameters and analysis of variance (one-way ANOVA) or Kruskal-Wallis tests for quantitative parameters, as appropriate.
Implementation of NIV | 01.06.2016-10.07.2018
  Is NIV implemented electively or urgently (yes versus no), in an outpatient or input setting (yes vs no), by liberal pulmonologist or hospital center (yes vs no). Data with binary outcome. All data were analyzed using descriptive statistics. Qualitative parameters were described as frequencies and percentages and quantitative parameters were described as mean and standard deviation (SD) or as median and interval interquartile (IQR). Comparisons between groups were performed using chi-square tests or Fisher exact tests for qualitative parameters and analysis of variance (one-way ANOVA) or Kruskal-Wallis tests for quantitative parameters, as appropriate.
Follow-up modalities | 01.06.2016-10.07.2018
  Arterial blood gas (ABG): pH, pCO2 (kPa), pO2 (kPa), HCO3 (mmol/l), base excess (mmol/l), SpO2 (%), spirometry: FEV1/FVC % of predicted, FEV1 % of predicted, FVC % of predicted, pulsoxicapnometry: SpO2 (%), time with SpO2 < 90% (%), desaturation index > 3 (%), pCO2 (kPa). All data were analyzed using descriptive statistics. Qualitative parameters were described as frequencies and percentages and quantitative parameters were described as mean and standard deviation (SD) or as median and interval interquartile (IQR). Comparisons between groups were performed using chi-square tests or Fisher exact tests for qualitative parameters and analysis of variance (one-way ANOVA) or Kruskal-Wallis tests for quantitative parameters, as appropriate.
Ventilators | 01.06.2016-10.07.2018
  Home ventilators used (ASV vs barometric vs volumetric), settings: minimal and maximal pressure support (cmH2O), fixed EPAP (cmH20), minimal and maximal EPAP (cmH2O), back-up respiratory rate (cycles/min), data downloaded from the device software: EPAP (cmH2O), IPAP (cmH2O), EPAP 90% (cmH2O), mean pressure support (cmH2O), tidal volume (ml), minute ventilation (L/min), leaks (L/min), apnea index (N/hour), apnea-hypopnea index (N/hour), mean daily use (min/day), interfaces (facial vs nasal vs prongs masks), duration to therapy (expressed in hours). All data were analyzed using descriptive statistics. Qualitative parameters were described as frequencies and percentages and quantitative parameters were described as mean and standard deviation (SD) or as median and interval interquartile (IQR).
Prevalence of home non invasive ventilation (NIV) | 01.06.2016-10.07.2018
  Prevalence of home non invasive ventilation. All data were analyzed using descriptive statistics. Qualitative parameters were described as frequencies and percentages and quantitative parameters were described as mean and standard deviation (SD) or as median and interval interquartile (IQR). Comparisons between groups were performed using chi-square tests or Fisher exact tests for qualitative parameters and analysis of variance (one-way ANOVA) or Kruskal-Wallis tests for quantitative parameters, as appropriate.
Barometric and volumetric ventilation versus adaptive servo-ventilation (ASV) | 01.06.2016-10.07.2018
  Sub-analysis groups depending on the type of home NIV (barometric and volumetric ventilation versus ASV). All data were analyzed using descriptive statistics. Qualitative parameters were described as frequencies and percentages and quantitative parameters were described as mean and standard deviation (SD) or as median and interval interquartile (IQR). Comparisons between groups were performed using chi-square tests or Fisher exact tests for qualitative parameters and analysis of variance (one-way ANOVA) or Kruskal-Wallis tests for quantitative parameters, as appropriate.
Medical follow-up | 01.06.2016-10.07.2018
  To study if there is a statistical significance in the outcomes listed above (diagnostic groups, comorbidities) depending if the medical follow-up is done by a liberal pulmonologist or a hospital center. All data were analyzed using descriptive statistics. Qualitative parameters were described as frequencies and percentages and quantitative parameters were described as mean and standard deviation (SD) or as median and interval interquartile (IQR). Comparisons between groups were performed using chi-square tests or Fisher exact tests for qualitative parameters and analysis of variance (one-way ANOVA) or Kruskal-Wallis tests for quantitative parameters, as appropriate.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Janssens JP, Derivaz S, Breitenstein E, De Muralt B, Fitting JW, Chevrolet JC, Rochat T. Changing patterns in long-term noninvasive ventilation: a 7-year prospective study in the Geneva Lake area. Chest. 2003 Jan;123(1):67-79. doi: 10.1378/chest.123.1.67. PMID 12527605
- [Derived] Cantero C, Adler D, Pasquina P, Uldry C, Egger B, Prella M, Younossian AB, Poncet A, Soccal-Gasche P, Pepin JL, Janssens JP. Adaptive Servo-Ventilation: A Comprehensive Descriptive Study in the Geneva Lake Area. Front Med (Lausanne). 2020 Apr 3;7:105. doi: 10.3389/fmed.2020.00105. eCollection 2020. PMID 32309284
- [Derived] Cantero C, Adler D, Pasquina P, Uldry C, Egger B, Prella M, Younossian AB, Soccal PM, Pepin JL, Janssens JP. Long-Term Noninvasive Ventilation in the Geneva Lake Area: Indications, Prevalence, and Modalities. Chest. 2020 Jul;158(1):279-291. doi: 10.1016/j.chest.2020.02.064. Epub 2020 Mar 31. PMID 32243941